CLINICAL TRIAL: NCT00862342
Title: Efficacy and Safety of Second-line Combination Chemotherapy With Avastin in Patients With Metastatic Colorectal Cancer Who Have Received First-line Chemotherapy Plus Avastin
Brief Title: Post-First Progression Use of Bevacizumab in Metastatic Colorectal Cancer (mCRC)
Acronym: SAFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae Won Kim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-2008-0487
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab continuation plus chemotherapy in patients who have failed previous bevacizumab plus other chemotherapy
  Interventions: Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — Bevacizumab plus chemotherapy (chemotherapy will be chosen by physician's decision)

SUMMARY:
Bevacizumab beyond progression has been proven to be safe in the community setting (BRiTE) and in the post-marketing study (BEAT), and confirmed its efficacy and safety in the first line with all regimens of chemotherapy. A total of 1,953 patients were treated in BRiTE. At median follow-up of 17.5 mo, there were 1,369 1st PD and 839 deaths. Among patients with 1st PD, 65.2% received any 2nd-line chemotherapy, 34.8% received cetuximab, and 53.8% received BBP. In a multivariate analysis, Bevacizumab beyond first progression and exposure to any 2nd-line chemotherapy were independently associated with increased overall survival (both p < 0.0001). Bevacizumab beyond progression appears to be associated with longer overall in BRiTE.

The investigators planned a prospective study to prove this phenomenon of bevacizumab beyond progression.

DETAILED DESCRIPTION:
Patients should have been treated with bevacizumab plus chemotherapy as a 1st line treatment, and after 1st progression, these patients will be accrued in this study of bevacizumab plus chemotherapy as a 2nd line treatment, and the combined chemotherapy will be chosen by physician's decision in consider with previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented colorectal adenocarcinoma
* Progression during first-line bevacizumab containing chemotherapy within 3 months
* No serious toxicity to bevacizumab of 1st line treatment
* Unresectable metastases
* Uni-dimensional measurable lesion(s) by RECIST
* Age over 18 years old
* ECOG 0-2
* Adequate organ functions by clinical laboratory exams

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* CNS metastases
* GI bleeding
* Hypersensitivity to any of chemotherapeutic agents
* Prior use of cetuximab or other targeted agents other than bevacizumab
* Major surgery within 6 weeks
* Other serious illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6 weeks

SECONDARY OUTCOMES:
Overall survival | 6 weeks
Toxicity profiles | 2 or 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, M.D., Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Result] Hong YS, Lee J, Kim KP, Lee JL, Park YS, Park JO, Park SH, Kim SY, Baek JY, Kim JH, Lee KW, Kim TY, Kim TW. Multicenter phase II study of second-line bevacizumab plus doublet combination chemotherapy in patients with metastatic colorectal cancer progressed after upfront bevacizumab plus doublet combination chemotherapy. Invest New Drugs. 2013 Feb;31(1):183-91. doi: 10.1007/s10637-012-9853-3. Epub 2012 Jul 11. PMID 22782485